CLINICAL TRIAL: NCT01122563
Title: Reproducibility Study of OABSS and Its Response to Treatment in Indonesia - Part 2: Responsiveness
Brief Title: A Study to Evaluate Response of Overactive Bladder Symptom Score (OABSS) to Treatment
Acronym: RESORT-2
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Indonesia Inc. (Industry)
Responsible Party: Disclosure Director, Astellas Pharma, Inc
Other Study IDs: EQL-CRU.005-2009
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Overactive Bladder
Keywords: OABSS; IPSS; PPBC; 3-day micturition diary; Solifenacin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Solifenacin — oral
  Other Names: Vesicare

SUMMARY:
This study is to evaluate change of overactive bladder symptom scores (OABSS) between, before and after solifenacin treatment to OAB subjects.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms OAB for 3 months or longer
* At least 3 urgency episode in last 3 days
* Symptoms of OAB as verified by the screening 3-day bladder diary, defined by:

  * Number of micturition ≥8 times/day
  * Number of urgency episodes in 3 days ≥3

Exclusion Criteria:

* Significant stress incontinence or mixed stress/urge incontinence
* Subject with indwelling catheters or practicing intermittent self-catheterization
* Symptomatic urinary tract infection, chronic inflammation
* Diabetic neuropathy
* Subjects who are prohibited from taking solifenacin as contraindications
* Drug or non-drug treatment for OAB was started, quitted or changed in 4 weeks
* Participation in any clinical trial in 30 days except for Part-1 of RESORT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic OAB patients having urgency episodes
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
OABSS | Weeks 0, 4 and 12

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | Weeks 0, 4 and 12
Quality of Life (QOL) Score | Weeks 0, 4 and 12
Patient Perception of Bladder Condition (PPBC) | Weeks 0, 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Indonesia
Locations (3):
- Indonesia (3):
  - Bandung
  - Jakarta
  - Surabaya